CLINICAL TRIAL: NCT04191226
Title: Overall Perspective on the Characteristics of Genetic Mutation in Recurrent Cervical Cancer
Brief Title: Genetic Mutation in Recurrent Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: CC-TMB
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Recurrent Cervical Cancer; Nucleotide Variant; Copy Number Variation; Insertion-deletion Variation; Genomic Structural Variation; Total Mutation Burden; Microsatellite Instability; PD-1; PD-L1
MeSH Terms: conditions — Uterine Cervical Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and paired tumor tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multi-gene panel testing — A multi-gene panel, which consists of more than 500 hundred genes will be provided for mutation analysis

SUMMARY:
Little is known about the characteristics of genetic mutation in recurrent cervical cancer. This study is to explore the targeted genetic mutations via a multi-gene panel, which consists of more than 500 hundred genes. The mutation characteristics are to be revealed in single nucleotide variants, copy number variations, insertion-deletion variations, and genomic structural variations. The total mutation burden (TMB) will be calculated. The status of microsatellite instability, expression of PD-1 and PD-L1 antibodies are also tested. These findings will be studies in association with the patients' prognosis and sensitivity to platinum-based chemotherapy and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Pathology confirmed of recurrent cervical adenocarcinoma, squamous carcinoma or adenosquamous carcinoma
* With available materials for analysis
* With detailed clinicopathological information
* Given consent to participate the trial

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of pathology confirmed of recurrent cervical adenocarcinoma, squamous carcinoma or adenosquamous carcinoma, and aged 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of genetic mutations | Two years
  Frequency of various genetic mutations among recruited patients

SECONDARY OUTCOMES:
Total mutation burden | Two years
  Total mutation burden calculated in definite patient
Frequency of microsatellite Instability | Two years
  Microsatellite Instability in definite patient
Expression rates of PD-1 and PD-L1 antibodies | Two years
  Expression rates of PD-1 and PD-L1 antibodies among recruited patients

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided